CLINICAL TRIAL: NCT04013555
Title: The Effects of Kynurenine Aminotransferase Inhibition in People With Schizophrenia
Acronym: TrypNAC-II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HP-00086009
Record Dates: First submitted 2019-06-27; First posted 2019-07-09 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Acetylcysteine; Tryptophan

STUDY DESIGN:
Intervention Model Description: This will be a double-blind, placebo-controlled, randomized cross-over challenge study. Participant randomization will use a permuted block randomization system (block sizes 2 or 4), in which treatment assignment order is random within each block, with an equal number of participants assigned to each treatment, to generate a list of treatment assignments. Thus, it will be difficult to ascertain the next treatment assignment, even if a participant becomes unblinded, while any imbalance in the number of participants between the treatment groups will be kept within tight limits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All raters, investigators and other staff will be blind to treatment assignment except for the research pharmacist. The research pharmacist does not participate in assessing any of the primary symptom or side effect dependent variables and conveys no information about treatment assignment to participants or staff except in a medical emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- N-acetylcysteine & Tryptophan (Experimental): N-acetylcysteine 140 mg/kg up to a maximum of 15 g. Thirty minutes after N-acetylcysteine administration participants will receive Tryptophan, 6 grams.
  Interventions: Drug: N-acetylcysteine (NAC); Drug: Tryptophan
- Placebo & Tryptophan (Placebo Comparator): Placebo 140 mg/kg up to a maximum of 15 g. Thirty minutes after placebo administration participants will receive Tryptophan, 6 grams.
  Interventions: Drug: Placebo; Drug: Tryptophan

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — Flavored effervescent formulation
  Other Names: Cetylev
  Arms: N-acetylcysteine & Tryptophan
Drug: Placebo — Flavored effervescent formulation designed to mimic NAC
  Arms: Placebo & Tryptophan
Drug: Tryptophan — Oral slurry form

SUMMARY:
Kynurenic acid (KYNA) is a naturally occurring chemical in the brain. Studies with rodents indicate that levels of KYNA can impact levels of the neurotransmitters glutamate and dopamine. One way to reliably increase KYNA levels is by ingesting the amino acid tryptophan. Tryptophan is a normal part of the human diet. Tryptophan gets metabolized/changed to other chemicals in the body- including KYNA. By giving people 6 grams of tryptophan, the investigators will be able to increase the KYNA level in a controlled way. The investigators will then be able to study the effects of KYNA on neurotransmitters by using cognitive tests and magnetic resonance imaging techniques (measuring brain activity and brain chemistry using the MRI magnet).

The overall goal of the study is to examine how the medication N-acetylcysteine (NAC), when added to tryptophan, affects various cognitive functions, such as verbal and visual memory. The investigators will also use magnetic resonance imaging (MRI) to examine how NAC affects brain activity and chemicals.

DETAILED DESCRIPTION:
The purpose of the study is to examine whether high dose N-acetylcysteine (NAC) blocks the adverse effects of increased kynurenic acid (KYNA) on selected measures of brain chemistry, function and behavior, through the inhibition of kynurenine aminotransferase (KAT) II, which converts kynurenine to KYNA. The study will be a double-blind, placebo-controlled, randomized cross-over challenge study, in which people with schizophrenia are pretreated with either high-dose NAC, 140 mg/kg up to a maximum of 15 g, or placebo, then receive tryptophan (TRYP), 6 gms. The tryptophan challenge method robustly increases peripheral measures of kynurenine and KYNA in humans and putatively increases brain KYNA levels, through the CNS conversion of kynurenine to KYNA; a process that is observed in both rodents and nonhuman primates. The investigators will evaluate the ability of NAC to inhibit the conversion of kynurenine to KYNA with the following primary outcome measures: 1) the investigators will measure serum kynurenine and KYNA before and after NAC/placebo pre-treatment and TRYP administration and examine whether NAC compared to placebo blocks the peripheral conversion of kynurenine to KYNA; 2) the investigators will use the arterial spin labeling (ASL) technique to measure whole brain and frontal gray matter cerebral blood flow (CBF) before and after NAC/placebo pre-treatment and TRYP administration and examine whether NAC compared to placebo attenuates the effects of TRYP on ASL CBF measures; 3) the investigators will use magnetic resonance spectroscopy (MRS) to measure glutamate and glutathione levels in the medial prefrontal cortex (mPFC) before and after NAC/placebo pre-treatment and TRYP administration and examine whether NAC compared to placebo increases MRS glutathione and glutamate measures; and 4) the investigators will use diffusion tensor imaging (DTI) to measure white matter fractional anisotropy (FA) before and after NAC/placebo pre-treatment and TRYP administration and examine whether NAC compared to placebo increases white matter FA.

The investigators will have two secondary endpoints. First, if the investigators observe that NAC attenuates the effects of TRYP on ASL and/or increases mPFC glutamate levels or white matter DTI FA, then the investigators will examine whether these effects are related to changes in cognitive measures of attention, verbal and visual memory, and working memory. Second, the investigators will use measures of serum KYNA and peripheral blood mononuclear cell (PBMC) kynurenine 3-monooxygenase (KMO) activity levels to examine whether the level of these measures is related to the observed effects of NAC on our neuroimaging and cognitive outcome measures.

The investigators hypothesize that NAC will inhibit KAT II, which will be reflected in the: 1) decreased peripheral conversion of kynurenine to KYNA; and 2) increased CBF, glutamate, and white matter fractional anisotropy (FA). In addition, the investigators hypothesize that the NAC effects on the neuroimaging measures will be related to improved performance on cognitive measures of attention, verbal and visual memory and working memory. These observed effects of NAC will be greater than those seen with placebo. The investigators further hypothesize that the NAC effects on ASL CBF, glutamate, and FA measures will be independent of NAC-induced changes in MRS glutathione, i.e., not due to the NAC oxidative stress mechanism, but, rather, will be correlated with NAC-induced reductions in the peripheral conversion of kynurenine to KYNA. Finally, the investigators hypothesize that the observed effects of NAC on CBF, glutamate, and FA will be related to baseline serum KMO activity and KYNA levels. The demonstration that NAC reverses the adverse impact of increased KYNA levels will importantly support the development of KAT II inhibitors for the enhancement of cognition in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age: 18 to 55 years
* DSM-5 Criteria for schizophrenia, schizoaffective disorder or schizophreniform disorder (documented by SCID)
* Prescription of antipsychotic medication for at least 60 days and constant dose for 30 days prior to study entry (either first or second generation antipsychotics permitted)
* Female participants must agree to use a medically accepted means of contraception

Exclusion Criteria:

* DSM-5 alcohol or substance misuse disorder in the last 3 months (documented by SCID)
* History of an organic brain disorder; mental retardation; or a medical condition, whose pathology or treatment could alter cognition
* Active disorders that have been reported to affect tryptophan metabolism or interfere with absorption will be excluded (Acute Intermittent Porphyria, Celiac Disease, Crohn's Disease, Irritable Bowel Syndrome; Brune and Pflughaupt 1975; Torres et al 2007).
* Excessive self-reported daily caffeine intake, defined as intake exceeding 1000mg or the equivalent of 8 cups of coffee
* Pregnancy or lactation
* No metal in body that will interfere with MR imaging
* Monoamine oxidase inhibitors, migraine headache medications (triptans) and dextromethorphan
* Forensic or legal issues

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, M.D., Principal Investigator — University of Maryland
Locations (1):
- Maryland Psychiatric Research Center (MPRC) ; the Treatment Research Program (TRP), Catonsville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-eight people were screened and consented for study participation. Fourteen participants were excluded and 4 were withdrawn prior to randomization. Seventy people were randomized.
Groups:
- N-acetylcysteine, Then Placebo: On Challenge Day 1, participants first received N-acetylcysteine, 140 mg/kg up to a maximum of 15 g. Thirty minutes after N-acetylcysteine administration participants received Tryptophan, 6 grams.
  On Challenge Day 2 (at least two weeks after Challenge Day #1), participants first received placebo, 140 mg/kg up to a maximum of 15 g. Thirty minutes after placebo administration participants received Tryptophan, 6 grams.
  N-acetylcysteine (NAC): Flavored effervescent formulation
  Placebo: Flavored effervescent formulation designed to mimic N-acetylcysteine.
  Tryptophan: Oral slurry form
- Placebo, Then N-acetylcysteine: On Challenge Day #1, participants first received placebo, 140 mg/kg up to a maximum of 15 g. Thirty minutes after placebo administration participants received Tryptophan, 6 grams.
  On Challenge Day #2 (at least 2 weeks after Challenge Day #1), participants first received N-acetylcysteine, 140 mg.kg up to a maximum of 15g. Thirty minutes after placebo administration participants received Tryptophan, 6 grams.
  N-acetylcysteine (NAC): Flavored effervescent formulation
  Placebo: Flavored effervescent formulation designed to mimic N-acetylcysteine.
  Tryptophan: Oral slurry form
Period: Challenge Day #1
Arm/Group | N-acetylcysteine, Then Placebo | Placebo, Then N-acetylcysteine
Started | 36 | 34
Completed | 29 | 29
Not Completed | 7 | 5
Period: Challenge Day #2
Arm/Group | N-acetylcysteine, Then Placebo | Placebo, Then N-acetylcysteine
Started (One of the participants randomized to the N-acetylcysteine, then placebo sequence dropped out of the study between the first and second challenge day.) | 28 | 29
Completed | 25 | 26
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: Participants randomized
Groups:
- N-acetylcysteine, Then Placebo: On Challenge Day 1, participants first received N-acetylcysteine, 140 mg/kg up to a maximum of 15 g. Thirty minutes after N-acetylcysteine administration participants received Tryptophan, 6 grams.
  On Challenge Day 2 (at least two weeks after Challenge Day #1), participants first received placebo, 140 mg/kg up to a maximum of 15 g. Thirty minutes after placebo administration participants received Tryptophan, 6 grams.
- Placebo, Then N-acetylcysteine: On Challenge Day #1, participants first received placebo, 140 mg/kg up to a maximum of 15 g. Thirty minutes after placebo administration participants received Tryptophan, 6 grams.
  On Challenge Day #2 (at least 2 weeks after Challenge Day #1), participants first received N-acetylcysteine, 140 mg.kg up to a maximum of 15g. Thirty minutes after placebo administration participants received Tryptophan, 6 grams.
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine, Then Placebo | Placebo, Then N-acetylcysteine | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 26 | 24 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 16 | 16 | 32
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Serum Kynurenine Levels
Description: The investigators will use the kynurenine serum measures to examine whether NAC compared to placebo blocks the peripheral conversion of kynurenine to KYNA.
Time Frame: Baseline, 1 hour and 4 hours on each Challenge Day
Population: Participants who completed at least one Challenge Day
Measure: Mean (Standard Deviation); unit: pmoles/ul
Arm/Group | N-acetylcysteine & Tryptophan | Placebo & Tryptophan
Number analyzed (Participants) | 54 | 54
pmoles/ul
  Baseline: number analyzed (Participants) | 54 | 53
  Baseline | 2.39 (1.89) | 1.97 (1.22)
  1 hour: number analyzed (Participants) | 51 | 54
  1 hour | 22.0 (18.4) | 23.3 (37.3)
  4 hours: number analyzed (Participants) | 52 | 52
  4 hours | 65.8 (51.6) | 94.0 (159.5)
Statistical Analysis 1: Comparison: N-acetylcysteine & Tryptophan vs Placebo & Tryptophan; Test type: Superiority; p < 0.05, Mixed Models Analysis; difference in difference = -12.78, Standard Error of Mean 6.33

2. Primary Outcome: Kynurenic Acid Levels
Description: The investigators will use the KYNA serum measures to examine whether NAC compared to placebo blocks the peripheral conversion of kynurenine to KYNA.
Time Frame: Baseline, 1 hour and 4 hours on each Challenge Day
Population: Participants who completed at least one Challenge Day
Measure: Mean (Standard Deviation); unit: fmoles/ul
Arm/Group | N-acetylcysteine & Tryptophan | Placebo & Tryptophan
Number analyzed (Participants) | 54 | 54
fmoles/ul
  Baseline: number analyzed (Participants) | 54 | 53
  Baseline | 48.1 (50.9) | 42.9 (35.2)
  1 hour: number analyzed (Participants) | 53 | 54
  1 hour | 1687 (3463) | 1322 (3382)
  4 hours: number analyzed (Participants) | 52 | 52
  4 hours | 5758 (4850) | 7471 (6930)
Statistical Analysis 1: Comparison: N-acetylcysteine & Tryptophan vs Placebo & Tryptophan; Test type: Superiority; p < 0.05, Mixed Models Analysis; difference in difference = -1766.8, Standard Error of Mean 550.7

3. Primary Outcome: Whole Brain Gray Matter Cerebral Blood Flow (CBF)
Description: The investigators will use a Pseudo-continuous Arterial Spin Labeling (pCASL) sequence, which provides full brain coverage with high spatial resolution and excellent WM signal-to-noise ratio (SNR) (SNR>15), to measure whole brain gray matter cerebral blood flow (CBF). The investigators will use the pCASL CBF measures to examine whether NAC compared to placebo attenuates the effects of TRYP on ASL CBF measures.
Time Frame: Baseline, 2 hours on each Challenge Day
Population: Participants who completed at least one Challenge Day
Measure: Mean (Standard Deviation); unit: ml/100 g/min
Arm/Group | N-acetylcysteine & Tryptophan | Placebo & Tryptophan
Number analyzed (Participants) | 53 | 54
ml/100 g/min
  Baseline | 49.9 (11.0) | 52.5 (10.3)
  2 hours | 54.4 (12.0) | 57.3 (12.2)
Statistical Analysis 1: Comparison: N-acetylcysteine & Tryptophan vs Placebo & Tryptophan; Test type: Superiority; p < 0.05, Mixed Models Analysis; difference in difference = -2.58, Standard Error of Mean 1.42

ADVERSE EVENTS:
Time Frame: Over 4 study visits (over 6-8 weeks)
Arm/Group | N-acetylcysteine & Tryptophan | Placebo & Tryptophan
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 2/63 | 2/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | N-acetylcysteine & Tryptophan (N=63) | Placebo & Tryptophan (N=64)
Nausea (Gastrointestinal disorders) | 2 | 2/29
Vomiting (Gastrointestinal disorders) | 2 | 2/29
Dizziness (Ear and labyrinth disorders) | 1 | 2/29
Anxiety (Psychiatric disorders) | 0 | 1/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT04013555/Prot_SAP_000.pdf